CLINICAL TRIAL: NCT02705560
Title: Randomized, Controlled, Cross-Over Study to Assess Dietary Biomarkers and Metabolic Effects After a Single Dose of Milk and Cheese in Healthy Subjects
Brief Title: Assessment of Dietary Biomarkers and Metabolic Effects After the Intake of Milk and Cheese
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Agroscope Liebefeld-Posieux Research Station ALP (Other)
Responsible Party: Principal Investigator, Francois Pralong, Prof, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 347/15
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — CD36 Antigens; Hardness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cow´s milk (3.9% fat, pasteurized) (Experimental): Cow´s milk (3.9% fat, pasteurized) Single dose, 600 ml milk
  Interventions: Other: Cow´s milk (3.9% fat, pasteurized)
- Hard, yellow cheese (Experimental): Hard, yellow cheese Single dose, 100 g cheese
  + 500 ml water
  Interventions: Other: hard, yellow cheese
- Soy based drink (Active Comparator): Soy based drink Single dose, 600 ml soy drink (soy drink + plant based cream)
  Interventions: Other: Soy based drink

INTERVENTIONS:
Other: Cow´s milk (3.9% fat, pasteurized) — 600 ml full fat milk (organic, pasteurized, 400 kcal)
  Arms: Cow´s milk (3.9% fat, pasteurized)
Other: hard, yellow cheese — 100 g Swiss cheese (Le Gruyère medium ripe, 400 kcal)
  Arms: Hard, yellow cheese
Other: Soy based drink — 600 ml Soy drink (540 ml soy milk (232 kcal) supplemented with 60 ml soy and plant based cream (167 kcal)
  Arms: Soy based drink

SUMMARY:
Dietary biomarkers are compounds in biofluids that directly reflect the intake of specific foods or food groups. Their exploration and use in the field of dietary assessments could provide an objective measure of actual intake complementing classical assessment methods (e.g. food frequency questionnaire, 24h recalls). To date, only a limited number of foods have been covered by validated biomarkers.

The study is part of the international project "The Food Biomarker Alliance (FOODBALL)". The study described here has been assigned to assess biomarkers of the intake of milk and cheese. Up to now, there is an evident lack of data on specific and validated biomarkers of milk and cheese (dairy products), which belong to the most relevant public health related foods in Europe. This study will further provide novel insights into the influence of fermentation of milk-based foods on metabolic effects and postprandial adaptations, which has not yet been studied in depth before using cheese as fermented product. Outcomes will support and expand earlier findings on correlation between the intake of fermented dairy products intake and human health.

DETAILED DESCRIPTION:
This is an acute, randomized, controlled, cross-over study designed to identify dietary biomarkers of milk and cheese intake and to asses metabolic effects after the ingestion of a non-fermented product (milk) and a fermented product (cheese) in healthy subjects.

Twelve healthy participants (six women, six men) in fasted state will consume three different foods in a randomized order on three different study days. Two days prior to each dietary intervention, the run-in period is initiated, during which participants have to follow a restricted diet. Participants will receive a standardised meal for the last dinner during run-in phase. The same meal will be served on the day of the dietary intervention for lunch and for dinner (period of controlled diet). Before and after ingestion of the test foods, blood samples and urine samples will be collected (up to 6 hours). Additionally, 24h-samples will be collected. Primary outcomes (metabolites) will be measured in blood serum and plasma collected at 6 different time points and in urine collected at 7 different time points. Transcriptomics analysis will be performed on whole blood samples collected at 4 time points while clinical chemistry parameters will be assessed in blood samples withdrawn at 6 different time points.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Aged 18 - 40 years
* BMI > 18.5 and < 30 kg/m2
* Daily consumption of milk
* No adverse effects after intake of 600 ml of milk

Exclusion Criteria:

* Smokers
* Diagnosed health condition (chronic or infectious disease)
* Taking medication (oral contraceptive pill is allowed)
* Taking nutritional supplements (e.g. vitamins, minerals)
* Pregnant, lactating
* Antibiotics treatment 6 months prior to intervention
* Allergy to milk
* Allergy to soy
* Known intolerance to lactose
* Other food allergies or intolerances (e.g. histamine)
* Anemia (hemoglobin < 120 g/l) at the screening visit
* Iron deficiency (ferritin < 30 µg/l) at the screening visit
* Not willing/able to consume all test foods (milk, cheese and soy drink)
* Not willing/able to consume standardized meals
* Not willing to avoid drinking alcohol during study days
* Not willing to follow nutritional restrictions during study days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-06 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Identification of dietary biomarkers of cheese and milk intake | 24 hours

SECONDARY OUTCOMES:
Transcriptomics analyses / gene expression | 6 hours
Blood cell count and cell type determination | 6 hours
Glucose | 24 hours
Insulin | 24 hours
Triacylglycerides | 24 hours
Total cholesterol | 24 hours
HDL cholesterol | 24 hours
LDL cholesterol | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: François Pralong, MD, Principal Investigator — CHUV
Locations (1):
- Service of Endocrinology, Diabetes and Metabolism, University Hospital, CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Pimentel G, Burnand D, Munger LH, Pralong FP, Vionnet N, Portmann R, Vergeres G. Identification of Milk and Cheese Intake Biomarkers in Healthy Adults Reveals High Interindividual Variability of Lewis System-Related Oligosaccharides. J Nutr. 2020 May 1;150(5):1058-1067. doi: 10.1093/jn/nxaa029. PMID 32133503
- [Derived] Munger LH, Trimigno A, Picone G, Freiburghaus C, Pimentel G, Burton KJ, Pralong FP, Vionnet N, Capozzi F, Badertscher R, Vergeres G. Identification of Urinary Food Intake Biomarkers for Milk, Cheese, and Soy-Based Drink by Untargeted GC-MS and NMR in Healthy Humans. J Proteome Res. 2017 Sep 1;16(9):3321-3335. doi: 10.1021/acs.jproteome.7b00319. Epub 2017 Aug 10. PMID 28753012